CLINICAL TRIAL: NCT03396835
Title: Desaturation Validation of INVSENSOR00009
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-19029
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- INVSENSOR00009 Sensor (Experimental): All subjects who are enrolled into the test group and participate in data collection receive both the INVSENSOR00009 and the control sensor simultaneously on the forehead.
  Interventions: Device: INVSENSOR00009

INTERVENTIONS:
Device: INVSENSOR00009 — All subjects who are enrolled into the test group and participate in data collection receive both the INVSENSOR00009 and the control sensor simultaneously on the forehead.

SUMMARY:
This study is designed to measure the trending accuracy of a noninvasive measurement of cerebral oxygen saturation. One Large sensor (adult sensor) and one INVSENSOR00009 will be placed on the subject's forehead. The values obtained by the INVSENSOR00009 will be compared to the values collected with the adult sensor.Data will be collected from healthy adult subjects while undergoing a desaturation procedure wherein the concentration of oxygen inhaled is slowly reduced until the subject's arterial oxygen saturation is approximately 70%. The subject will then be returned to inhaling room air.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-50 years of age.
* Subject weighs a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall.
* Hemoglobin value is greater than or equal to 11 g/dL.
* Baseline heart rate ≥ 45 bpm and ≤ 85 bpm.
* Carbon monoxide (CO) value ≤ 2.0% FCOHb (Fractional saturation of hemoglobin with Carbon monoxide)
* Subject has a physical status of American Society of Anesthesiology (ASA) I or II (American Society of Anesthesiology Class I; Healthy subjects without any systemic disease at all. American Society of Anesthesiology Class II; subjects with mild systemic disease) as it applies to the systemic disease portion of the classification.
* Systolic Blood Pressure ≤ 140 mmHg and Diastolic Blood Pressure ≤ 90 mmHg.
* Subject is able to read and communicate in English and understands the study and risks involved.

Exclusion Criteria:

* Subject is pregnant.
* Subject smokes (smoking includes e-cigarette use).
* Subject has a BMI > 35 and has been classified as morbidly obese or at an increased risk for participation by a medical professional.
* Subject has open wounds, inflamed tattoos or piercings, visible healing wounds.
* Subject experiences frequent or severe headaches and/or migraine headaches.
* Subject has known drug or alcohol abuse and/or use of recreational drugs.
* Subject has experienced a concussion or head injury with loss of consciousness within the last year.
* Subject has any chronic bleeding disorders (i.e. hemophilia).
* Subject has any history of a stroke, myocardial infarction, seizures or heart attack.
* Subject has any cancer or history of cancer (not including skin cancer).
* Subject has a chronic neurological disease (i.e. multiple sclerosis, Huntington's Disease).
* Subject has any cardiac dysrhythmia(s) (i.e. atrial fibrillation) and has not received clearance by their physician to participate.
* Subject has a known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder) that interferes with the subject's level of consciousness.
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study (Discretion of investigator).
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome.
* Subject who has taken anticoagulant medication within the last 30 days.
* Subject has taken opioid pain medication within 24 hours of start of study.
* Subject has either signs or history of peripheral ischemia.
* Subject has had invasive surgery within the past year- including but not limited to major dental surgery, gallbladder, heart, appendix, major fracture repairs (involving plates/ screws), jaw surgery, urinary tract surgery, plastic surgery, major ear nose and throat (ENT) surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery.
* Subject has donated blood within the past 30 days.
* Subject has symptoms of congestion, head colds, flu or other illnesses.
* Subject experiences claustrophobia or has generalized anxiety disorder.
* Subject has been in severe car accident(s) or a similar type of accident(s) requiring hospitalization within the last 12 months.
* Subject has chronic unresolved asthma, lung disease or respiratory disease.
* Subject is allergic to lidocaine, latex, adhesives, or plastic.
* Subject has heart conditions, insulin-dependent diabetes or uncontrolled hypertension.
* Subject has given vaginal delivery, had a pregnancy terminated, a miscarriage with hospitalization, or had a C-section within the last 6 months.
* Discretion of investigator/study staff.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Clinical Lab, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00009 Sensor
Started | 16
Completed | 14
Not Completed | 2
Not completed — Withdrawn prior to completion | 1
Not completed — Did not meet criteria for data analysis | 1

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00009 Sensor
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants] — Population: One subject was withdrawn prior to completing study procedures. One subject did not meet criteria for data analysis.
  Participants
    number analyzed (Participants) | 14
    <=18 years | 0
    Between 18 and 65 years | 14
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject was withdrawn prior to completing study procedures. One subject did not meet criteria for data analysis.
  Participants
    number analyzed (Participants) | 14
    Female | 7
    Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One subject was withdrawn prior to completing study procedures. One subject did not meet criteria for data analysis.
  Participants
    White: number analyzed (Participants) | 14
    White | 4
    Hispanic: number analyzed (Participants) | 14
    Hispanic | 3
    Asian or Pacific Islander: number analyzed (Participants) | 14
    Asian or Pacific Islander | 1
    African American: number analyzed (Participants) | 14
    African American | 6
Region of Enrollment [Count of Participants; unit: Participants] — Population: One subject was withdrawn prior to completing study procedures. One subject did not meet criteria for data analysis.
  Participants
    United States: number analyzed (Participants) | 14
    United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Trending Regional Oxygen Saturation Accuracy of the INVSENSOR00009 Relative to the Control Sensor by Arms Calculation
Description: Trending ARMs accuracy is defined as root mean squared relative error of all data points of all subjects. Accuracy of the sensors will be determined by comparing regional oxygen saturation (rSO2) readings from INVSENSOR00009 and control sensor and calculating the Arithmetic root mean square (ARMS) value.
Time Frame: 1-5 hours
Measure: Number; unit: % tissue oxygen saturation
Arm/Group | INVSENSOR00009 Sensor
Number analyzed (Participants) | 14
% tissue oxygen saturation | 1.3

ADVERSE EVENTS:
Time Frame: 1 to 5 hours
Arm/Group | INVSENSOR00009 Sensor
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT03396835/Prot_SAP_000.pdf